CLINICAL TRIAL: NCT07101601
Title: An Open-label, Dose-finding, Phase 1 Study to Assess the Safety, Tolerability, Efficacy, and Pharmacokinetic Profile, and to Explore the Pharmacodynamic Profile of DM5167 in Patients With Advanced Solid Tumors
Brief Title: Study of DM5167 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: DIGMBIO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DM001-101
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1: Dose-escalation Cohort 1 (Experimental): The first level of dose of DM5167
  Interventions: Drug: DM5167
- Part 1: Dose-escalation Cohort 2 (Experimental): The second level of dose of DM5167
  Interventions: Drug: DM5167
- Part 1: Dose-escalation Cohort 3 (Experimental): The third level of dose of DM5167
  Interventions: Drug: DM5167
- Part 1: Dose-escalation Cohort 4 (Experimental): The fourth level of dose of DM5167
  Interventions: Drug: DM5167
- Part 1: Dose-escalation Cohort 5 (Experimental): The fifth level of dose of DM5167
  Interventions: Drug: DM5167
- Part 1: Dose-escalation Cohort 6 (Experimental): The sixth level of dose of DM5167
  Interventions: Drug: DM5167
- Part 2: Dose-expansion Cohort (Experimental): The recommended Phase 2 dose of DM5167
  Interventions: Drug: DM5167

INTERVENTIONS:
Drug: DM5167 — Once daily for 28 days

SUMMARY:
DM5167 is a second-generation of PARP inhibitor that selectively targets the PARP-1 enzyme. This results in less haematological toxicity and a high level of safety.

The aim of the study is to assess the safety and tolerability of DM5167 in patients with advanced solid tumors not respond to other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 19 years or older as of the date of written informed consent
* Patients who have at least one measurable lesion according to RECIST version 1.1
* ECOG performance status ≤ 1
* Patients with life expectancy ≥ 12 weeks
* Patients who meet the clinical laboratory test criteria confirming adequate liver, renal, and hematologic function
* Patients who voluntarily provide written informed consent to participate in this study
* Patients with histologically or cytologically confirmed unresectable advanced solid tumors
* Patients who have BRCA1/BRCA2 mutations

Exclusion Criteria:

* Patients with a medical history of significant illness
* Patients with QT interval of > 450 ms (for men) or > 460 ms (for women)\
* Patients who have not yet recovered from toxicity related to previous anticancer therapy
* Patients were predicted to demonstrate hypersensitivity to the components of the investigational medicinal product
* Patients who have participated in another clinical trial and received an investigational product or medical device
* Other individuals deemed inappropriate for participation in the study by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of dose limiting toxicities (DLT) of DM5167 | During the first cycle (28 days) of DM5167 treatment
  Determined by National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) version 5.0
Part 1 and Part 2: Treatment emergent adverse events (TEAE) and serious adverse events (SAEs) | First dose up to 28 days post end of treatment
  Clinically significant changes in vital signs, physical examination, ECG and clinical laboratory tests graded by NCI CTCAE v5.0

SECONDARY OUTCOMES:
Area Under Curve (AUC) of DM5167 | - Cycle 1 - Day 1 & Day 15: pre-dose (0h) and up to 24 h post administration of DM5167 - Cycle 3, 5, 7 - Day 1: pre-dose
  AUC from the time of dosing to the time of the last measurable concentration
Objective response rate (ORR) | Through study completion, an average of 1 year
  The proportion of subjects with best overall response (BOR) evaluated by RECIST version 1.1
Maximum Concentration (Cmax) of DM5167 | - Cycle 1 - Day 1 & Day 15: pre-dose (0h) and up to 24 h post administration of DM5167 - Cycle 3, 5, 7 - Day 1: pre-dose
  Maximum observed concentration after administration

OTHER OUTCOMES:
PARP inhibition in blood | Cycle 1, 2, 3, 5, 7 - Day 1: before the administration of DM5167
  Change in poly (ADP-ribose) (PAR) levels in peripheral blood mononuclear cells (PBMCs))

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient privacy, confidentiality, and compliance with applicable data protection regulations.